CLINICAL TRIAL: NCT06045975
Title: Durvalumab/Tremelimumab in Neoadjuvant and Adjuvant Setting in Patients With HCC Treated by by Percutaneous Ablation Procedure in Curative Intent: French Multicenter Phase 2 Therapeutic
Brief Title: Durvalumab/Tremelimumab in Neoadjuvant and Adjuvant Setting in Patients With HCC Treated by by Percutaneous Ablation Procedure
Acronym: DUMELEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP220729
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: HCC; Electroporation; immunotherapy; radiofrequency ablation; microwave
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab/Tremelimumab (Experimental): Durvalumab/Tremelimumab in neoadjuvant and Durvalumab in adjuvant setting
  Interventions: Drug: Durvalumab/Tremelimumab in neoadjuvant and Durvalumab in adjuvant setting

INTERVENTIONS:
Drug: Durvalumab/Tremelimumab in neoadjuvant and Durvalumab in adjuvant setting — * Durvalumab 1500 mg/Tremelimumab 300 mg infusion in a neoadjuvant setting followed by PA procedure at Day 30+/-7 days
  * 11 monthly Durvalumab 1500 mg infusions.

SUMMARY:
This project is a Phase 2 trial testing the safety and efficacy of treatment with Durvalumab/Tremelimumab in neoadjuvant and Durvalumab in adjuvant setting in patients with BCLC A HCC treated by by percutaneous ablation (PA) procedure in a curative intent.

DUMELEP is a Multicentre, Phase 2 trial

Eligible patients will receive consecutively:

1. 1 Durvalumab 1500 mg/Tremelimumab 300 mg infusion in a neoadjuvant setting
2. percutaneous ablation procedure in a curative attempt at Day 30
3. 11 monthly Durvalumab 1500 mg infusions.
4. Classical follow-up during an additional year (every 3 months)

DETAILED DESCRIPTION:
Immunotherapy is currently the gold standard for first-line treatment of advanced HCC based of the combination of check-point inhibitors (CPI). The first approved regimen is based on the association of atezolizumab and bevacizumab, an antiangiogenic molecule. More recently, the HIMALAYA trial demonstrated the superiority of durvalumab-tremelimumab over sorafenib, establishing a new first-line option.The combination of Immunotherapy and locoregional treatments in earlier HCC stages may reduce relapse rates. Preliminary data from the IMBRAVE 050 trail reports lower rates of recurrence following HCC percutaneous ablation (PA) or resection associated with atezolizumab and bevacizumab in adjuvant setting.PA procedures and most likely electroporation induce T-cell recruitment that may foster immunomodulation. In particular, radiofrequency ablation (RFA) can lead to stimulation of NK cells with a more differentiated and proactivatory phenotypic profile with general increase of functional activities. As compared with RFA, these local changes of IRE induce more robust systemic effects, including both tumorigenic and immunogenic events. Indeed, the preservation of the tumor microvasculature and extracellular matrix within the coagulated zone would favour infiltration by anti tumoral immune cells. These observations are relevant for development of neoadjuvant and adjuvant immunotherapeutic strategies in the setting of HCC treated by percutaneous ablation, and particularly IRE .

Neoadjuvant and adjuvant trials using these new molecules must now be cautiously designed based on the rigorous selection of special populations and therapeutic indications based on the following criteria:

* Exclusion of early forms of HCC with low probability of recurrence for statistical power issues
* Inclusion of patients with HCC treated in "curative intent" by new PA techniques such as electroporation
* Selective inclusion of patients treated with PA whose immunomodulatory properties are recognized

ELIGIBILITY:
Inclusion criteria

* Male or female patients ≥ 18 years of age
* Histological or radiological diagnosis of HCC
* Patients with newly diagnosed or recurrent HCC (following a previous curative procedure performed at least 6 months before inclusion) eligible for PA as assessed by multidisciplinary board corresponding to BCLC A stage:
* Uninodular HCC ≥ 2 cm and ≤ 5 cm, no macroscopic vascular invasion
* Multinodular maximum 3 nodules ≤ 3 cm
* Body weight >30 kg
* Liver function status Child-Pugh Class A
* <<Eastern Cooperative Oncology Group (ECOG)>><<World Health Organisation (WHO) performance status of 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory tests:
* Total bilirubin ≤ 2 mg/dL
* Serum creatinine ≤ 1.5 x ULN
* Lipase ≤ 2 x ULN
* Prothrombine time-international normalized ratio (PT-INR) < 2.3 and PTT < 1.5
* Glomerular Filtration Rate (GFR) ≥ 30 mL/min/1.73 m2
* Life expectancy ≥ 3 months
* Women of childbearing potential (WOCBP) need to accept one effective method of contraception until 3 months after the last infusion of durvalumab and avoid pregnancy
* Patients affiliated to a Social Security System
* Written informed consent signed (patients must be free from tutelle, curatelle or sauvegarde de justice)
* Haemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC ≥1.0 × 109/L)
* Platelet count ≥75 × 109/L
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.)
* AST (SGOT) and ALT (SGPT) ≤5x ULN
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patients must have a life expectancy of at least 12 weeks
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at pre inclusion/inclusion. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to inclusion
* Patients infected with HCV must be managed according to international recommendations
* Antiviral therapy in case of HBV active infection or inactive carriage

Non inclusion criteria

* Patients with contraindications to PA procedure (Pacemakers or patients who have a history of cardiac arrhythmias or irregular heartbeats in case of IRE, ascites, Coagulopathy, Ongoing infection)
* Patients with contraindication to contrast medium intravenous injection either gadolinium or iodinate
* Prior liver transplantation
* Uncontrolled HCC defined by the absence of remission > 6months following resection of percutaneous ablation at time of inclusion
* Prior systemic treatment for HCC, in particular agents targeting T-cell costimulation or checkpoint pathways (including those targeting PD-1, PD-L1 or PD-L2, CD137, or cytotoxic Tlymphocyte antigen [CTLA-4]).
* Patients with uncontrolled HBV infection and viral load above 100 IU/mL.
* Patients with large esophageal varices at risk of bleeding that are not being treated with conventional medical intervention
* Past or concurrent history of neoplasm other than HCC, except for in situ carcinoma of the cervix uteri and/or non-melanoma skin cancer and superficial bladder tumors. Any cancer curatively treated > 3 years prior to study entry is permitted
* Major surgical procedure or significant traumatic injury within 28 days before enrolment
* Congestive heart failure New York Heart Association (NYHA) ≥ class 2
* Unstable angina or myocardial infarction within the past 6 months before enrolment
* Grade 3 (severe) hypertension ≥180 and/or ≥110 mmHG (systolic and diastolic, according to National Heart Foundation 2016)
* Patients with phaeochromocytoma
* Refractory ascites according to EASL guidelines definition (ascites that cannot be mobilized or the early recurrence of which cannot be prevented because of a lack of response to sodium restriction and diuretic treatment)
* Persistent proteinuria of NCI-CTCAE version 5.0 ≥ Grade 3
* Ongoing infection > Grade 2 according to NCI-CTCAE version 5.0.
* Patients with chronic hepatitis B or inactive carriers for HBV must be under anti-HBV treatment
* Clinically significant bleeding NCI-CTCAE version 5.0 ≥ Grade 3 within 30 days before enrolment
* Any psychological, familial, sociological, geographical or illness or medical condition that could jeopardize the safety of the patient and/or his compliance with the study protocol and follow-up procedure
* Known history of human immunodeficiency virus (HIV) infection
* Non-healing wound, ulcer or bone fracture
* Known hypersensitivity to the study drug or excipients in the formulation
* Any malabsorption condition
* Breast feeding
* Pregnancy
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab and tremelimumab combination therapy.
* Participation in another clinical study with an investigational product during the last 6 months
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria :

  1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.

Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable. <<amend as required based on any combination studies with other anticancer agents>>

* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for :

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Study excludes patients with -brain metastases or spinal cord compression: Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry. Brain metastases will not be recorded as RECIST Target Lesions at baseline if study allows patients with brain metastases.
* Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging (RECIST)) for details on the imaging modality) obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases.

These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent <<and anti-convulsants>> for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.

* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
* History of active primary immunodeficiency
* Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab and tremelimumab combination therapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Patients who have received prior anti-PD-1, anti-PD-L1 or anti-CTLA-4:

  1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
  3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
  4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2028-09-28 (Estimated)

PRIMARY OUTCOMES:
local recurrence-free survival | 12 months after PA procedure
  Local recurrence is defined as the emergence of irregular areas enhanced at arterial phase followed by wash out at portal phase observed next to the ablation zone

SECONDARY OUTCOMES:
Changes of tumorous and non-tumorous perfusion parameters | one month of neoadjuvant treatment
  rates of nodule(s) comprising necrosis and/or hypoperfusion radiological aspect compared before and after neoadjuvant course): analyzed as qualitative variables
Changes of size of nodules following neoadjuvant course | one month of neoadjuvant treatment
  Nodule rates of early response after a single procedure of PA procedure (defined as absence of active tumor evaluated at one month following PA procedure)
Incidences of intra segmental/ extra segmental distant recurrence | Throughout the study, an average of 30 months
  will be assessed using imaging techniques as recommended by international guidelines (3-months US and MRI)
Overall survival | 12 months after PA procedure
  defined as patients who are alive with or without HCC recurrence 1 year after PA procedure. Causes of death will be specified when applicable during this timeframe.
Overall survival | 12 months after PA procedure
  defined as patients who are alive with or without HCC recurrence 1 year after PA procedure. Date of death will be specified when applicable during this timeframe.
Treatment-related adverse events | Throughout the study, an average of 30 months
  will be monitored according to manufacturer guidelines and recommendation.
Timeframe of PA performance | one month of neoadjuvant treatment
  defined as number of days of delay in case of safety issues encountered
Compliance to neoadjuvant and adjuvant treatments | during one cycle neoadjuvant treatment and 11 months starting after the PA evaluation
  Respect of scheduled Durvalumab/Tremelimumab infusions, Number of Durvalumab/Tremelimumab infusions administered
Safety of Durvalumab/Tremelimumab infusions | Throughout the study, an average of 30 months
  Incidence of Adverse Events using current CTCAE

OTHER OUTCOMES:
Assessment of tumour architecture and cytology : Histological outcome measures | From inclusion to PA procedure; assessed up to 30 days
  Absence of tumour cells (binary scale :0/1)
Assessment of tumour architecture and cytology : Histological outcome measures | From inclusion to PA procedure; assessed up to 30 days
  Assessment of intra and extra tumoral inflammatory infiltrate (semi quantitative scale: 0=non, 1=mild, 2=intense)
Assessment of tumour architecture and cytology :Genomics | From inclusion to PA procedure; assessed up to 30 days
  Change in gene expression following sequential whole exome sequencing (binary scale 0/1 with clustering analyses)
Absence of tumour cells (binary scale: 0/1) | At inclusion, and at the time of the PA procedure
  Consittution of a sequential biobank comprising liver tissue : histological outcome
Assessment of intra and extra tumoral inflammatory infiltrate (semi quantitative scale: 0=non, 1=mild, 2=intense) outcome | At inclusion, and at the time of the PA procedure
  Consittution of a sequential biobank comprising liver tissue : histological
Consittution of a sequential biobank comprising liver tissue : Genomics | At inclusion, and at the time of the PA procedure
  hange in gene expression following sequential whole exome sequencing (binary scale 0/1 with clustering analyses)
Consittution of a sequential biobank comprising peripheral samples (serum, plasma) | At inclusion,at EP procedure ; at 1, 3, 6, 9 and 11 months after PA procedure
  Changes in PIGF (UI/mL), VEGF-A (UI/mL), VEGF-C (UI/mL), sVEGFR2 (UI/mL), sVEGFR3 (UI/mL), MET (UI/mL), sKIT (UI/mL), Ang2 (UI/mL), AFP (UI/mL), PIVKA (UI/mL) (changes expressed by median comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Perre NAHON, MD-PhD, Principal Investigator — APHP
Locations (1):
- Hospitl Avicenne, Bobigny, France

REFERENCES:
- [Background] Trinchet JC, Bourcier V, Chaffaut C, Ait Ahmed M, Allam S, Marcellin P, Guyader D, Pol S, Larrey D, De Ledinghen V, Ouzan D, Zoulim F, Roulot D, Tran A, Bronowicki JP, Zarski JP, Goria O, Cales P, Peron JM, Alric L, Bourliere M, Mathurin P, Blanc JF, Abergel A, Serfaty L, Mallat A, Grange JD, Buffet C, Bacq Y, Wartelle C, Dao T, Benhamou Y, Pilette C, Silvain C, Christidis C, Capron D, Thiefin G, Hillaire S, Di Martino V, Nahon P, Chevret S; ANRS CO12 CirVir Group. Complications and competing risks of death in compensated viral cirrhosis (ANRS CO12 CirVir prospective cohort). Hepatology. 2015 Sep;62(3):737-50. doi: 10.1002/hep.27743. Epub 2015 Mar 20. PMID 25678021
- [Background] N'Kontchou G, Mahamoudi A, Aout M, Ganne-Carrie N, Grando V, Coderc E, Vicaut E, Trinchet JC, Sellier N, Beaugrand M, Seror O. Radiofrequency ablation of hepatocellular carcinoma: long-term results and prognostic factors in 235 Western patients with cirrhosis. Hepatology. 2009 Nov;50(5):1475-83. doi: 10.1002/hep.23181. PMID 19731239
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] Seror O. Ablative therapies: Advantages and disadvantages of radiofrequency, cryotherapy, microwave and electroporation methods, or how to choose the right method for an individual patient? Diagn Interv Imaging. 2015 Jun;96(6):617-24. doi: 10.1016/j.diii.2015.04.007. Epub 2015 May 14. PMID 25981214
- [Background] Seror O, N'Kontchou G, Ibraheem M, Ajavon Y, Barrucand C, Ganne N, Coderc E, Trinchet JC, Beaugrand M, Sellier N. Large (>or=5.0-cm) HCCs: multipolar RF ablation with three internally cooled bipolar electrodes--initial experience in 26 patients. Radiology. 2008 Jul;248(1):288-96. doi: 10.1148/radiol.2481071101. Epub 2008 May 15. PMID 18483229
- [Background] Sutter O, Calvo J, N'Kontchou G, Nault JC, Ourabia R, Nahon P, Ganne-Carrie N, Bourcier V, Zentar N, Bouhafs F, Sellier N, Diallo A, Seror O. Safety and Efficacy of Irreversible Electroporation for the Treatment of Hepatocellular Carcinoma Not Amenable to Thermal Ablation Techniques: A Retrospective Single-Center Case Series. Radiology. 2017 Sep;284(3):877-886. doi: 10.1148/radiol.2017161413. Epub 2017 Apr 28. PMID 28453431
- [Background] Cheng RG, Bhattacharya R, Yeh MM, Padia SA. Irreversible Electroporation Can Effectively Ablate Hepatocellular Carcinoma to Complete Pathologic Necrosis. J Vasc Interv Radiol. 2015 Aug;26(8):1184-8. doi: 10.1016/j.jvir.2015.05.014. Epub 2015 Jun 26. PMID 26119204
- [Background] Niessen C, Beyer LP, Haimerl M, Schicho A, Stroszczynski C, Wiggermann P, Jung EM. Percutaneous irreversible electroporation of hepatocellular carcinoma: Contrast-enhanced ultrasound-findings during 1-year follow-up. Clin Hemorheol Microcirc. 2019;72(1):85-93. doi: 10.3233/CH-180449. PMID 30584122
- [Background] Niessen C, Beyer LP, Pregler B, Dollinger M, Trabold B, Schlitt HJ, Jung EM, Stroszczynski C, Wiggermann P. Percutaneous Ablation of Hepatic Tumors Using Irreversible Electroporation: A Prospective Safety and Midterm Efficacy Study in 34 Patients. J Vasc Interv Radiol. 2016 Apr;27(4):480-6. doi: 10.1016/j.jvir.2015.12.025. Epub 2016 Feb 26. PMID 26922979
- [Background] Niessen C, Thumann S, Beyer L, Pregler B, Kramer J, Lang S, Teufel A, Jung EM, Stroszczynski C, Wiggermann P. Percutaneous Irreversible Electroporation: Long-term survival analysis of 71 patients with inoperable malignant hepatic tumors. Sci Rep. 2017 Mar 7;7:43687. doi: 10.1038/srep43687. PMID 28266600
- [Background] Bhutiani N, Philips P, Scoggins CR, McMasters KM, Potts MH, Martin RC. Evaluation of tolerability and efficacy of irreversible electroporation (IRE) in treatment of Child-Pugh B (7/8) hepatocellular carcinoma (HCC). HPB (Oxford). 2016 Jul;18(7):593-9. doi: 10.1016/j.hpb.2016.03.609. Epub 2016 May 1. PMID 27346140
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Behm B, Di Fazio P, Michl P, Neureiter D, Kemmerling R, Hahn EG, Strobel D, Gress T, Schuppan D, Wissniowski TT. Additive antitumour response to the rabbit VX2 hepatoma by combined radio frequency ablation and toll like receptor 9 stimulation. Gut. 2016 Jan;65(1):134-43. doi: 10.1136/gutjnl-2014-308286. Epub 2014 Dec 18. PMID 25524262
- [Background] Zerbini A, Pilli M, Laccabue D, Pelosi G, Molinari A, Negri E, Cerioni S, Fagnoni F, Soliani P, Ferrari C, Missale G. Radiofrequency thermal ablation for hepatocellular carcinoma stimulates autologous NK-cell response. Gastroenterology. 2010 May;138(5):1931-42. doi: 10.1053/j.gastro.2009.12.051. Epub 2010 Jan 11. PMID 20060829
- [Background] Bulvik BE, Rozenblum N, Gourevich S, Ahmed M, Andriyanov AV, Galun E, Goldberg SN. Irreversible Electroporation versus Radiofrequency Ablation: A Comparison of Local and Systemic Effects in a Small-Animal Model. Radiology. 2016 Aug;280(2):413-24. doi: 10.1148/radiol.2015151166. Epub 2016 Jan 27. PMID 27429143
- [Background] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Background] Iida N, Nakamoto Y, Baba T, Nakagawa H, Mizukoshi E, Naito M, Mukaida N, Kaneko S. Antitumor effect after radiofrequency ablation of murine hepatoma is augmented by an active variant of CC Chemokine ligand 3/macrophage inflammatory protein-1alpha. Cancer Res. 2010 Aug 15;70(16):6556-65. doi: 10.1158/0008-5472.CAN-10-0096. Epub 2010 Jul 27. PMID 20663902
- [Background] Kelley RK, Sangro B, Harris W, Ikeda M, Okusaka T, Kang YK, Qin S, Tai DW, Lim HY, Yau T, Yong WP, Cheng AL, Gasbarrini A, Damian S, Bruix J, Borad M, Bendell J, Kim TY, Standifer N, He P, Makowsky M, Negro A, Kudo M, Abou-Alfa GK. Safety, Efficacy, and Pharmacodynamics of Tremelimumab Plus Durvalumab for Patients With Unresectable Hepatocellular Carcinoma: Randomized Expansion of a Phase I/II Study. J Clin Oncol. 2021 Sep 20;39(27):2991-3001. doi: 10.1200/JCO.20.03555. Epub 2021 Jul 22. PMID 34292792
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Abou-Alfa GK, Lau G, Kudo M, Chan SL, Kelley RK, Furuse J, Sukeepaisarnjaroen W, Kang YK, Van Dao T, De Toni EN, Rimassa L, Breder V, Vasilyev A, Heurgue A, Tam VC, Mody K, Thungappa SC, Ostapenko Y, Yau T, Azevedo S, Varela M, Cheng AL, Qin S, Galle PR, Ali S, Marcovitz M, Makowsky M, He P, Kurland JF, Negro A, Sangro B. Tremelimumab plus Durvalumab in Unresectable Hepatocellular Carcinoma. NEJM Evid. 2022 Aug;1(8):EVIDoa2100070. doi: 10.1056/EVIDoa2100070. Epub 2022 Jun 6. PMID 38319892